CLINICAL TRIAL: NCT05605158
Title: Comparative Clinical Study to Evaluate the Possible Beneficial Effect of Empagliflozin Versus Pioglitazone on Non-diabetic Patients With Non-Alcoholic Steatohepatitis
Brief Title: Comparative Clinical Study Between Empagliflozin Versus Pioglitazone in Non-diabetic Patients With Non-alcoholic Steatohepatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Khaled Mohammed Elnawasany, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35937/10/22
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Non Alcoholic Steatohepatitis
Keywords: NASH; Nonalcoholic fatty liver disease (NAFLD); SGLT2i; Empagliflozin; Pioglitazone; Hepatic steatosis index (HSI); Fibrosis index based on the 4 factors (FIB-4); Aspartate transaminase-to-platelet ratio index (APRI); Cytokeratin-18; Transforming growth factor-beta1 (TGF-β1); Malondialdehyde (MDA)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Camurati-Engelmann Syndrome | interventions — Pioglitazone; empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Pioglitazone group; n=28) (Active Comparator): Non-diabetic patients with non-alcoholic steatohepatitis will receive 30mg/day pioglitazone for 24 weeks.
  Interventions: Drug: Pioglitazone 30mg
- Group 2 (Empagliflozin group; n=28) (Active Comparator): Non-diabetic patients with non-alcoholic steatohepatitis will receive 10mg/day empagliflozin for 24 weeks.
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Pioglitazone 30mg — Pioglitazone 30 mg will be administered orally once daily for 24 weeks.
  Arms: Group 1 (Pioglitazone group; n=28)
Drug: Empagliflozin 10 MG — Empagliflozin 10 mg will be administered orally once daily for 24 weeks.
  Arms: Group 2 (Empagliflozin group; n=28)

SUMMARY:
This study aims to evaluate the possible beneficial effect of empagliflozin versus pioglitazone on non-diabetic patients with non-alcoholic steatohepatitis (NASH).

This study will be a randomized, comparative parallel study. The study will be conducted according to the ethical standards of Helsinki declaration in 1964 and its later amendments.

The study duration will be 24 weeks. The patients will be randomized into two groups:

Group 1: (Pioglitazone group; n=28) which will receive 30mg/day pioglitazone for 24 weeks.

Group 2: (Empagliflozin group; n=28) which will receive 10mg/day empagliflozin for 24 weeks.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a condition of fat accumulation in the liver in the absence of alcohol consumption. Dyslipidemia predominantly hypertriglyceridemia, oxidative stress and insulin resistance play crucial roles in the pathogenesis of NASH. Non-alcoholic fatty liver (NAFL) and non-alcoholic steatohepatitis (NASH) are the two major subtypes of NAFLD. The patients diagnosed with NASH can subsequently progress to liver fibrosis, which increases the risks of cirrhosis and liver cancer. In Egypt, the prevalence of NAFLD is rising owing to rising prevalence of obesity whereas NAFLD was diagnosed in 57.65% of a cohort of obese Egyptian adolescents. Furthermore, around 1 in 3 had steatosis, and 1 in 20 had moderate-to-advanced fibrosis in Egypt.

NASH is also associated with production of various atherogenic factors including pro-inflammatory cytokines such as tumor necrosis factor-α (TNF-α) which has been proposed to be the key link between obesity and insulin resistance during NASH. Current guidelines recommend changing lifestyle patterns as first-line therapy strategy for NAFLD. However, there is no defined treatment for NAFLD, previous studies aimed at discovering new treatments for NAFLD and several treatment approaches have been proposed, such as insulin-sensitizers, lipid-lowering drugs, antioxidants, L-carnitine, pentoxifylline, probiotics, ezetimibe, sitagliptin, empagliflozin, pentoxifylline, dapagliflozin, pioglitazone, and lobeglitazone which were reported to reduce liver fat and improve ALT levels in patients with NASH and NAFLD through their anti-inflammatory, antioxidant, and antifibrogenic effects.

Cytokeratin 18 (CK18) is an intermediate filament protein expressed by hepatocytes. Cytokeratin 18 is released into the blood by cell death and hepatocyte apoptosis. Transforming growth factor beta-1 (TGF-β1) cytokine mediates the transformation of quiescent hepatic stellate cells (HSCs) into myofibroblast-like cells with an increased production of extra cellular matrix proteins. TGF-β1 concentration is elevated in patients with NASH as compared to patients with hepatic steatosis, suggesting that this cytokine is involved in the fibrogenesis during NASH.

Although pioglitazone has been proven to enhance metabolism and liver histology among patients with NAFLD, it has limitations in clinical use due to significant adverse events including weight gain, lower extremity edema and risk for heart failure. Pioglitazone is a peroxisome proliferator activated receptor γ (PPARγ) agonist which can protect the liver by improving insulin resistance in patients with NAFLD and T2DM. It has been shown that pioglitazone could improve biochemical and histological parameters in non-diabetic patients with NASH. Previous trial revealed that, pioglitazone improved hepatic fibrosis in patients with NAFLD.

Sodium-glucose co-transporter type-2 inhibitors (SGLT2i) are glucose-lowering agents that improve glucose panel, promote weight loss and reduce serum uric acid level. There is increasing interest regarding the implication of SGLT2i in the treatment of NAFLD, regardless of the co-existence of T2DM. The beneficial effects of SGLT2i on NAFLD appear to be mediated directly through regulation of Endoplasmic Reticulum stress, oxidative stress, low-grade inflammation, autophagy and apoptosis. Empagliflozin (SGLT2i) was reported to decrease the expression of pro-fibrotic genes such as alpha smooth muscle actin (α-SMA), collagen, type I, alpha 1(collagen1α1), Matrix Metalloproteinase -2 (MMP2), and Transforming growth factor beta (TGF-β).

Furthermore, Empagliflozin successively induced the phosphorylation of MST1/2 and YAP, the two central members of the Hippo signaling pathway, in the CDAHFD-induced liver fibrosis leading to inhibition of HSCs activation and proliferation. In EFFECT-II trial, Dapagliflozin (SGLT2i) was found to reduce the levels of all measured hepatocyte injury biomarkers including cytokeratin 18-M30.

This study will be a randomized, comparative parallel study. The patients will be recruited from Outpatient Clinic of the Endocrine and Diabetes Unit, Tanta University Hospital, Tanta, Egypt. The diagnosis of NASH will be confirmed by imaging technique (increased liver echogenicity, stronger echoes in the hepatic parenchyma, vessel blurring, and narrowing of the lumen of the hepatic veins), mild to moderate elevation in aminotransferase activities (>2 but <5 times upper limit of normal), hepatic steatosis index (HSI) >36, HAIR score (hypertension, alanine aminotransferase level, insulin resistance) of 2 or 3. The study will be conducted according to the ethical standards of Helsinki declaration in 1964 and its later amendments. The study duration will be 24 weeks. The patients will be randomized into two groups:

Group 1: (Pioglitazone group; n=28) which will receive 30mg/day pioglitazone for 24 weeks.

Group 2: (Empagliflozin group; n=28) which will receive 10mg/day empagliflozin for 24 weeks.

* All patients will be submitted to demography, physical examination, and measurement of waist circumferences, weight, height, and calculation of body mass index (BMI).
* Ultrasonography of the liver will be carried out at baseline and at the end of the study.
* All patients will be assessed for complete blood count, glycated hemoglobin (HbA1c %), fasting blood glucose, fasting insulin, serum creatinine, liver panel, fasting lipid profile, serum Cytokeratin-18, serum transforming growth factor-beta1(TGF-β1), Malondialdehyde (MDA) and Tumor necrosis factor- alpha (TNF-α).
* The Homeostasis Model Assessment-insulin resistance (HOMA-IR), Hepatic steatosis index (HSI), HAIR score and Fibrosis risk scores including Fibrosis index based on the 4 factors (FIB-4) and Aspartate transaminase-to-platelet ratio index (APRI) will be calculated.
* All patients will be followed up by weekly telephone calls and monthly direct meetings according to scheduled visits to assess their adherence and to report any drug related adverse effects.

The primary outcome is the change in fibrosis indices (FIB-4 and APRI) and the liver enzymes. The secondary outcome is the change in measured biological markers mainly cytokeratin-18, MDA, TNF-α, and TGF-β1.

* Sample size calculation:

The sample size was calculated depending up-on a previous Randomized Controlled Trial included Fifty patients with NAFLD who were randomly assigned to either the empagliflozin group 10 mg daily or the control group (standard treatment without empagliflozin) for 20 weeks. The two groups showed a significant difference (P = 0.005) for the change in serum ALT level. In this context, the initial sample size of 50 patients will be sufficient to provide a good power to detect the effect. Assuming that, the attrition rate is 10%, the initial sample size will be 56 patients in both groups.

* Ethical approval:

The study will be conducted according to the ethical standards of Helsinki declaration in 1964 and its later amendments. The study will be approved by the Research Ethical Committee of Tanta University. The study will be registered as a clinical trial on clinicaltrial.gov. All participants will be informed about the benefits and risks of the study. Any unexpected risks that will appear during the course of the research will be clarified to the participants and to the ethical committee on time. The data of the enrolled patients will be confidential. All enrolled patients will give their written informed consents.

* Statistical analysis:

  1. The collected data will be tabulated using Microsoft® Office Excel, 2019 (Microsoft Corporation).
  2. The statistical analysis will be carried out using SPSS statistical package version 26.0 (IBM corporation software group, USA).
  3. Data will be tested for normality using Shapiro-Wilk test or Kolmogorov-Smirnov test.
  4. Parametric data will be analyzed using Paired and un-Paired t-test to compare the means within the same group and to compare the means of the two groups respectively.
  5. Non-parametric data will be analyzed using Mann Whitney U test to compare the means within the same group and to compare the means between groups.
  6. Categorical data will be analyzed using Chi-Square test.
  7. Fisher's exact test will be used to analyses the reported adverse effects.
  8. Correlation between variables will be assessed using Pearson or Spearman correlation coefficient which appropriate.
  9. Data will be expressed as the mean ±SD, medians, range, number and percent as appropriate.
  10. The significance level will be set at p≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic patients.
* Both males and females.
* Age >18 years old.
* Patient with body mass index (BMI) > 30 kg/m2.
* Patients with established diagnosis of NASH based on liver ultrasonography, mild to moderate elevation in aminotransferase activities (>2 but <5 times upper limit of normal), hepatic steatosis index (HSI) >36, and HAIR score of 2 or 3.

Exclusion Criteria:

* Patients with BMI > 40 kg/m2.
* Patients with type 2 diabetes mellitus (T2DM) on the basis of a fasting plasma glucose (FPG) level ≥ 126 mg/dl (7mmol/L) or glycated hemoglobin (HbA1c) > 6.5% (48 mmol/mol).
* Alcohol consumption greater than 20 g per day for women or greater than 30 g for men for at least three consecutive months over the past 5 years.
* History of viral hepatitis, hemochromatosis, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, biliary obstruction, alpha-1 antitrypsin deficiency.
* Patients on medications interfere with lipid and carbohydrate metabolisms.
* Patients with heart failure (New York Heart Association (NYHA) class 2-4).
* Patients with history of cardiovascular events within the past 3 months.
* Patients with renal impairment (eGFR> 45 mL/min/ 1.73 m2).
* Patients with cancer or with a history of cancer treatment over the past 2 years.
* Patients with thyroid disorder.
* Patients on medications associated with steatosis such as Non-steroidal anti-inflammatory drugs (NSAIDs), amiodarone, tamoxifen, estrogen, sodium valproate, corticosteroids, and methotrexate.
* Patients with inflammatory diseases.
* Patients on supplements known to have antioxidant activity such as vitamin E, vitamin C, zinc, and selenium.
* Pregnant and breastfeeding women.
* Females on oral contraceptive pills will be also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in fibrosis index based on the 4 factors (FIB-4) | Baseline and 24th week
  FIB-4 will be calculated using the formula: FIB-4 = Age (years)× AST (IU/L)/[platelet count (109/L) × ALT1/2 (IU/L)].
Change in aspartate transaminase-to-platelet ratio index (APRI) | Baseline and 24th week
  APRI will be calculated using the formula: APRI = (AST (IU/L)/upper limit of normal AST range) X 100 /platelet count (109/L).
Change in liver enzymes | Baseline, 12th and 24th week
  Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and Gamma-glutamyl transferase (GGT) will be determined by kinetic method.

SECONDARY OUTCOMES:
Cytokeratin-18 (CK-18) | Baseline and 24th week
  Serum level of cytokeratin-18 (CK-18) will be determined by Enzyme-linked Immunosorbent assay kits.
Malondialdehyde (MDA) | Baseline and 24th week
  Serum level of Malondialdehyde (MDA) will be assessed by colorimetric method.
Tumor necrosis factor-alpha (TNF-α) | Baseline and 24th week
  Serum levels of Tumor necrosis factor-alpha (TNF-α) will be determined by Enzyme-linked Immunosorbent assay kits.
Transforming growth factor-beta1 (TGF-β1) | Baseline and 24th week
  Serum levels of Transforming growth factor-beta1 (TGF-β1) will be determined by Enzyme-linked Immunosrbent assay kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Abenavoli L, Greco M, Milic N, Accattato F, Foti D, Gulletta E, Luzza F. Effect of Mediterranean Diet and Antioxidant Formulation in Non-Alcoholic Fatty Liver Disease: A Randomized Study. Nutrients. 2017 Aug 12;9(8):870. doi: 10.3390/nu9080870. PMID 28805669
- [Background] Abenavoli L, Milic N, Di Renzo L, Preveden T, Medic-Stojanoska M, De Lorenzo A. Metabolic aspects of adult patients with nonalcoholic fatty liver disease. World J Gastroenterol. 2016 Aug 21;22(31):7006-16. doi: 10.3748/wjg.v22.i31.7006. PMID 27610012
- [Background] Androutsakos T, Nasiri-Ansari N, Bakasis AD, Kyrou I, Efstathopoulos E, Randeva HS, Kassi E. SGLT-2 Inhibitors in NAFLD: Expanding Their Role beyond Diabetes and Cardioprotection. Int J Mol Sci. 2022 Mar 13;23(6):3107. doi: 10.3390/ijms23063107. PMID 35328527
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] El-Haggar SM, Mostafa TM. Comparative clinical study between the effect of fenofibrate alone and its combination with pentoxifylline on biochemical parameters and liver stiffness in patients with non-alcoholic fatty liver disease. Hepatol Int. 2015 Jul;9(3):471-9. doi: 10.1007/s12072-015-9633-1. Epub 2015 May 9. PMID 25956613
- [Background] Eriksson JW, Lundkvist P, Jansson PA, Johansson L, Kvarnstrom M, Moris L, Miliotis T, Forsberg GB, Riserus U, Lind L, Oscarsson J. Effects of dapagliflozin and n-3 carboxylic acids on non-alcoholic fatty liver disease in people with type 2 diabetes: a double-blind randomised placebo-controlled study. Diabetologia. 2018 Sep;61(9):1923-1934. doi: 10.1007/s00125-018-4675-2. Epub 2018 Jul 3. PMID 29971527
- [Background] Hasegawa T, Yoneda M, Nakamura K, Makino I, Terano A. Plasma transforming growth factor-beta1 level and efficacy of alpha-tocopherol in patients with non-alcoholic steatohepatitis: a pilot study. Aliment Pharmacol Ther. 2001 Oct;15(10):1667-72. doi: 10.1046/j.1365-2036.2001.01083.x. PMID 11564008
- [Background] Heo YJ, Lee N, Choi SE, Jeon JY, Han SJ, Kim DJ, Kang Y, Lee KW, Kim HJ. Empagliflozin Reduces the Progression of Hepatic Fibrosis in a Mouse Model and Inhibits the Activation of Hepatic Stellate Cells via the Hippo Signalling Pathway. Biomedicines. 2022 Apr 29;10(5):1032. doi: 10.3390/biomedicines10051032. PMID 35625768
- [Background] Kuchay MS, Krishan S, Mishra SK, Farooqui KJ, Singh MK, Wasir JS, Bansal B, Kaur P, Jevalikar G, Gill HK, Choudhary NS, Mithal A. Effect of Empagliflozin on Liver Fat in Patients With Type 2 Diabetes and Nonalcoholic Fatty Liver Disease: A Randomized Controlled Trial (E-LIFT Trial). Diabetes Care. 2018 Aug;41(8):1801-1808. doi: 10.2337/dc18-0165. Epub 2018 Jun 12. PMID 29895557
- [Background] Lee YH, Kim JH, Kim SR, Jin HY, Rhee EJ, Cho YM, Lee BW. Lobeglitazone, a Novel Thiazolidinedione, Improves Non-Alcoholic Fatty Liver Disease in Type 2 Diabetes: Its Efficacy and Predictive Factors Related to Responsiveness. J Korean Med Sci. 2017 Jan;32(1):60-69. doi: 10.3346/jkms.2017.32.1.60. PMID 27914133
- [Background] Lian J, Fu J. Pioglitazone for NAFLD Patients With Prediabetes or Type 2 Diabetes Mellitus: A Meta-Analysis. Front Endocrinol (Lausanne). 2021 Apr 28;12:615409. doi: 10.3389/fendo.2021.615409. eCollection 2021. PMID 33995271
- [Background] Lucero D, Zago V, Lopez GI, Graffigna M, Fainboim H, Miksztowicz V, Merono T, Belli S, Levalle O, Wikinski R, Brites F, Berg G, Schreier L. Pro-inflammatory and atherogenic circulating factors in non-alcoholic fatty liver disease associated to metabolic syndrome. Clin Chim Acta. 2011 Jan 14;412(1-2):143-7. doi: 10.1016/j.cca.2010.09.025. Epub 2010 Sep 29. PMID 20887718
- [Background] Machado MV, Cortez-Pinto H. Non-invasive diagnosis of non-alcoholic fatty liver disease. A critical appraisal. J Hepatol. 2013 May;58(5):1007-19. doi: 10.1016/j.jhep.2012.11.021. Epub 2012 Nov 23. PMID 23183525
- [Background] Powell EE, Wong VW, Rinella M. Non-alcoholic fatty liver disease. Lancet. 2021 Jun 5;397(10290):2212-2224. doi: 10.1016/S0140-6736(20)32511-3. Epub 2021 Apr 21. PMID 33894145
- [Background] Shimizu M, Suzuki K, Kato K, Jojima T, Iijima T, Murohisa T, Iijima M, Takekawa H, Usui I, Hiraishi H, Aso Y. Evaluation of the effects of dapagliflozin, a sodium-glucose co-transporter-2 inhibitor, on hepatic steatosis and fibrosis using transient elastography in patients with type 2 diabetes and non-alcoholic fatty liver disease. Diabetes Obes Metab. 2019 Feb;21(2):285-292. doi: 10.1111/dom.13520. Epub 2018 Oct 2. PMID 30178600
- [Background] Stefan N, Haring HU, Cusi K. Non-alcoholic fatty liver disease: causes, diagnosis, cardiometabolic consequences, and treatment strategies. Lancet Diabetes Endocrinol. 2019 Apr;7(4):313-324. doi: 10.1016/S2213-8587(18)30154-2. Epub 2018 Aug 30. PMID 30174213
- [Background] Sviklane L, Olmane E, Dzerve Z, Kupcs K, Pirags V, Sokolovska J. Fatty liver index and hepatic steatosis index for prediction of non-alcoholic fatty liver disease in type 1 diabetes. J Gastroenterol Hepatol. 2018 Jan;33(1):270-276. doi: 10.1111/jgh.13814. PMID 28464337
- [Background] Tomah S, Hamdy O, Abuelmagd MM, Hassan AH, Alkhouri N, Al-Badri MR, Gardner H, Eldib AH, Eid EA. Prevalence of and risk factors for non-alcoholic fatty liver disease (NAFLD) and fibrosis among young adults in Egypt. BMJ Open Gastroenterol. 2021 Oct;8(1):e000780. doi: 10.1136/bmjgast-2021-000780. PMID 34610926
- [Background] Zhang Y, Liu X, Zhang H, Wang X. Efficacy and Safety of Empagliflozin on Nonalcoholic Fatty Liver Disease: A Systematic Review and Meta-Analysis. Front Endocrinol (Lausanne). 2022 Feb 24;13:836455. doi: 10.3389/fendo.2022.836455. eCollection 2022. PMID 35282455